CLINICAL TRIAL: NCT00000391
Title: A Phase I Trial of Intranasal Peptide T: Safety, Toxicity, and Pharmacokinetics in Human Immunodeficiency Virus-1 (HIV-1) Infected Patients.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: 89 MH-SF
Record Dates: First submitted 2000-01-17; First posted 2000-01-18 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2002-04

CONDITIONS: HIV Infections
Keywords: Acquired Immunodeficiency Syndrome; AIDS-Related Complex
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Peptide T

INTERVENTIONS:
Drug: Peptide T

SUMMARY:
To study the safety and toxicity of intranasal peptide T (D-Ala-1-peptide-T-amide) in humans, and to find out how quickly and how much of a given dose enters the bloodstream and how quickly it leaves the bloodstream. To obtain information on the ability of intranasal peptide T to prevent, halt, and/or reverse the effects of AIDS on the central nervous system.

Studies have shown that AIDS is caused by a retrovirus. This virus works by inactivating or destroying human CD4 cells (which are part of the human immune system). This in turn leads to the observed immunologic defects and related illnesses, including HIV encephalopathy (disease of the brain). One method of preventing AIDS is to prevent HIV from entering the cell. HIV binds to the receptor CD4 site. Peptide T also binds to this site, and thus by competing for that site, can block the binding of the virus to its receptor. Preliminary animal and human studies indicate that peptide T is safe at the doses selected for this trial.

Thirty patients with AIDS or AIDS related complex (ARC) are entered into the study to receive an increasing schedule of three dosage levels of intranasal peptide T for 12 - 16 weeks followed by a 1-month off-drug follow-up period and a subsequent 1-month return to the drug. All patients receive an initial intravenous test dose of peptide T. The test dose is administered over 1 hour, followed by an observation period of 8 hours in the outpatient clinic.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have:

HIV infection. Ability to give informed consent. Ability to participate in an outpatient study.

* Allowed: Short course antimicrobials.
* Not breast-feeding
* Abstinence or agree to use barrier methods of birth control / contraception during the study
* Not pregnant
* Negative pregnancy test
* CD4 100 to 500 cells/mm3 (100 - 200 - 300 - 400 - 500).
* Creatinine > 1.6 mg/dl
* Hemoglobin >= 12 g/dl
* Platelet Count >= 100000 /mm3

Exclusion Criteria:

* Excluded: Asymptomatic HIV seropositive or lymphadenopathy syndrome diagnoses only (CDC criteria).
* Patients with the following conditions are excluded: Evidence of life-threatening opportunistic infection at time of entry into trial. Clinical evidence of active central nervous system disease secondary to immune dysregulation associated with HIV infection. Previous history of major psychiatric illness prior to 1977 or the time of initial exposure to HIV, if that is known. Evidence of clinically significant major psychiatric disturbance other than depression.
* Excluded within 4 weeks of study entry: Suramin. Antiretroviral agents. Anticancer treatments. Psychoactive agents.
* Excluded: Antivirals or immunomodulators.
* Excluded within 4 weeks of study entry: Radiation.
* Evidence of active substance abuse during 30 days prior to entry into trial. All behavior that can put patient at risk for reinfection with HIV: sexual contact with others known to have HIV infection, unsafe sexual practices, or sharing of needles or other intravenous equipment.
* Breast-feeding
* Positive pregnancy test
* Pregnant
* No abstinence or no agreement to use barrier methods of birth control / contraception during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 1988-01; Primary Completion 1990-01 (Actual)

PRIMARY OUTCOMES:
Radioimmunoassay for viral load | 12-16 weeks, 1 month
  The subsequent return to the drug for 1 month is after a 1 month off-drug follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Bridge TP, Study Chair — National Institute of Mental Health (NIMH)
Locations (1):
- Fenway Clinic, Boston, Massachusetts, United States